CLINICAL TRIAL: NCT04499677
Title: Favipiravir, Lopinavir/Ritonavir or Combination Therapy: a Randomised, Double Blind, 2x2 Factorial Placebo-controlled Trial of Early Antiviral Therapy in COVID-19
Brief Title: FLARE: Favipiravir +/- Lopinavir: A RCT of Early Antivirals
Acronym: FLARE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: LifeArc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 132084
Record Dates: First submitted 2020-06-16; First posted 2020-08-05 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2021-12

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — favipiravir; Lopinavir; lopinavir-ritonavir drug combination

STUDY DESIGN:
Intervention Model Description: Randomised, double-blind, 2x2 factorial placebo-controlled
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Favipiravir + Lopinavir/ritonavir (LPV/r) (Experimental): Oral favipiravir at 1800 mg twice daily on Day 1, followed by 400 mg four (4) times daily from Day 2 to Day 7 PLUS Lopinavir/ritonavir (LPV/r) at 400mg/100 mg twice daily on Day 1, followed by 200mg/50mg four (4) times daily from Day 2 to Day 7
  Interventions: Drug: Favipiravir; Drug: Lopinavir/ Ritonavir
- Favipiravir + Lopinavir/ritonavir (LPV/r) placebo (Experimental): Oral favipiravir at 1800 mg twice daily on Day 1, followed by 400 mg four (4) times daily from Day 2 to Day 7 PLUS Lopinavir/ritonavir (LPV/r) matched placebo at 400mg/100mg twice daily on Day 1, followed by 200mg/50mg four (4) times daily from Day 2 to Day 7.
  Interventions: Drug: Favipiravir; Other: Lopinavir/ Ritonavir Placebo
- Favipiravir placebo + Lopinavir/ritonavir (LPV/r) (Experimental): Oral favipiravir matched placebo at 1800 mg twice daily on Day 1, by 400 mg four (4) times daily from Day 2 to Day 7 PLUS Lopinavir/ritonavir (LPV/r) at 400mg/100mg twice daily on Day 1, followed by 200mg/50mg four (4) times daily from Day 2 to Day 7.
  Interventions: Drug: Lopinavir/ Ritonavir; Other: Favipiravir Placebo
- Favipiravir placebo + Lopinavir/ritonavir (LPV/r) placebo (Placebo Comparator): Oral favipiravir matched placebo at 1800 mg twice daily on Day 1, by 400 mg four (4) times daily from Day 2 to Day 7 PLUS Lopinavir/ritonavir (LPV/r) matched placebo at 400mg/100mg twice daily on Day 1, followed by 200mg/50mg four (4) times daily from Day 2 to Day 7.
  Interventions: Other: Favipiravir Placebo; Other: Lopinavir/ Ritonavir Placebo

INTERVENTIONS:
Drug: Favipiravir — Dosage and method of administration: Day 1: 1800 mg twice daily; Day 2 to Day 7: 400 mg four (4) times daily.
  Other Names: Avigan
  Arms: Favipiravir + Lopinavir/ritonavir (LPV/r); Favipiravir + Lopinavir/ritonavir (LPV/r) placebo
Drug: Lopinavir/ Ritonavir — Dosage and method of administration: Day 1: 400mg/100 mg twice daily; Day 2 to Day 7: 200mg/50mg four (4) times daily
  Other Names: Kaletra
  Arms: Favipiravir + Lopinavir/ritonavir (LPV/r); Favipiravir placebo + Lopinavir/ritonavir (LPV/r)
Other: Favipiravir Placebo — Dosage and method of administration: Day 1: 1800 mg twice daily; Day 2 to Day 7: 400 mg four (4) times daily.
  Arms: Favipiravir placebo + Lopinavir/ritonavir (LPV/r); Favipiravir placebo + Lopinavir/ritonavir (LPV/r) placebo
Other: Lopinavir/ Ritonavir Placebo — Dosage and method of administration: Day 1: 1800 mg twice daily; Day 2 to Day 7: 400 mg four (4) times daily.
  Arms: Favipiravir + Lopinavir/ritonavir (LPV/r) placebo; Favipiravir placebo + Lopinavir/ritonavir (LPV/r) placebo

SUMMARY:
The current pandemic of SARS-CoV-2 causing COVID-19 disease is an unprecedented global emergency. COVID-19 appears to be a disease with an early phase where the virus replicates, coinciding with first presentation of symptoms, followed by a later 'inflammatory' phase which results in severe disease in some individuals. It is known from other rapidly progressive infections such as sepsis and influenza that early treatment with antimicrobials is associated with better outcome. Antiviral medications are most likely to be effective when administered soon after infection. There is therefore an urgent need to study subjects who have recently developed symptoms, or have recently been tested positive with or without symptoms, and who can be sampled frequently to understand changes in viral load. This cohort will allow us to collect detailed trajectory data on early disease and understand how pharmacological interventions may affect this. The objective of the FLARE trial is to assess whether early antiviral therapy with either favipiravir + Lopinavir/ritonavir (LPV/r), LPV/r or favipiravir is associated with a decrease in viral load compared with placebo. The hypothesis is that this holds for COVID-19 and that early antiviral treatment may prevent progression to the later phase of the disease.

DETAILED DESCRIPTION:
FLARE is a phase IIA randomised, double-blind, 2x2 factorial placebo-controlled, interventional trial in which 240 participants, aged 18 years (≥ 18 years) to 70 years old inclusive will be recruited. Participants will be adults who have developed the early symptoms of COVID-19 within the first 5 days, or tested positive for SARS-CoV-2 within the first 7 days of symptom onset, or not presenting symptoms but tested positive within the last 48 hours (date/time of test must be within 48 hours of enrolment).

Eligible participants will be randomised 1:1:1:1 to receive one of the following combinations:

Favipiravir + Lopinavir/ritonavir (LPV/r) (both active); Favipiravir active + Lopinavir/ritonavir (LPV/r) placebo; Favipiravir placebo + Lopinavir/ritonavir (LPV/r) active; Favipiravir placebo + Lopinavir/ritonavir (LPV/r) placebo;

All participants will be enrolled and followed up for 28 days. A saliva sample for virological analysis and safety blood samples will be collected at baseline, as well as a diagnostic nose and throat swab, if the participant hasn't been tested for COVID-19 yet. Following randomisation, participants will take trial medication for 7 days and during this period will take a daily saliva sample and complete a symptoms diary including four daily temperature measurements.

Participants will have two follow-up visits at Day 7 and Day 14 where they will be assessed and undergo blood tests for toxicity and pharmacokinetic assessment (on Day 7 only) and provide stool samples. Participants will have a telephone follow up three (3) weeks after their last day of treatment (Day 7) and further information will be collected through a questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. Any adult with the following:

   * Symptoms compatible with COVID-19 disease (Fever >37.8oC on at least one occasion AND either cough and/ or anosmia) within the first 5 days of symptom onset
   * OR ANY symptoms compatible with COVID-19 disease (may include, but are not limited to fever, cough, shortness of breath, malaise, myalgia, headache, coryza) and tested positive for SARS-CoV-2 within the first 7 days of symptom onset
   * OR no symptoms but tested positive for SARS-CoV-2 within the last 48 hours (date/time of test must be within 48 hours of enrolment)
2. Male or female aged 18 years to 70 years old inclusive at screening
3. Willing and able to take daily saliva samples
4. Able to provide full informed consent and willing to comply with trial-related procedures

Exclusion Criteria:

1. Known hypersensitivity to any of the active ingredients or excipients in favipiravir and matched placebo, and in lopinavir/ritonavir and matched placebo
2. Chronic liver disease at screening (known cirrhosis of any aetiology, chronic hepatitis (e.g. autoimmune, viral, steatohepatitis), cholangitis or any known elevation of liver aminotransferases with AST or ALT > 3 X ULN)*
3. Chronic kidney disease (stage 3 or beyond) at screening: eGFR < 60 ml/min/1.73m2*
4. HIV infection, if untreated, detectable viral load or on protease inhibitor therapy
5. Any clinical condition which the investigator considers would make the participant unsuitable for the trial
6. Concomitant medications known to interact with favipiravir and matched placebo, and with lopinavir/ritonavir and matched placebo, and carry risk of toxicity for the participant
7. Current severe illness requiring hospitalisation
8. Pregnancy and/ or breastfeeding
9. Eligible female participants of childbearing potential and male participants with a partner of childbearing potential not willing to use highly effective contraceptive measures during the trial and within the time point specified following last trial treatment dose.
10. Participants enrolled in any other interventional drug or vaccine trial (co-enrolment in observational studies is acceptable).

    * Considering the importance of early treatment of COVID-19 to impact viral load, the absence of chronic liver/ kidney disease will be confirmed verbally by the participant during pre-screening and Screening/Baseline visit. Safety blood samples will be collected at Screening/Baseline visit (Day 1) and test results will be examined as soon as they become available within 24 hours.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2020-09-24 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-01-17 (Actual)

PRIMARY OUTCOMES:
Upper respiratory tract viral load at Day 5 | Day 5 from randomisation
  Quantitative polymerase chain reaction (PCR) performed on saliva samples at Day 5 of therapy

SECONDARY OUTCOMES:
Percentage of participants with undetectable upper respiratory tract viral load after 5 days of therapy | 5 days from randomisation
  Quantitative polymerase chain reaction (PCR) performed on saliva samples at Day 5 of therapy
Proportion of participants with undetectable stool viral load after 7 days of therapy. | 7 days from randomisation
  Quantitative polymerase chain reaction (PCR) performed on stool samples at Day 7
Rate of decrease in upper respiratory tract viral load during 7 days of therapy | 7 days
  PCR performed on daily saliva samples collected between Day 1 and Day 7 post-randomisation
Duration of fever following commencement of medication | 7 days
  Daily body temperature records between Day 1 and Day 7 post-randomisation
Proportion of participants with hepatotoxicity after 7 days of therapy | 7 days from randomisation
  Standard diagnostic laboratory assays for liver transaminases, alkaline phosphatase and bilirubin
Proportion of participants with other medication-related toxicity after 7 days of therapy and 14 days post-randomisation | Day 7 and Day 14 from randomisation
  Determination of medication-related adverse events by investigators at Day 7 and Day 14 post-randomisation
Proportion of participants admitted to hospital with COVID-19 related illness | 28 days
  Participant self-report, review of hospital records and discharge summaries within 28 days of randomisation
Proportion of participants admitted to ICU with COVID-19 related illness | 28 days
  Participant self-report, review of hospital records and discharge summaries within 28 days of randomisation
Proportion of participants who have died with COVID-19 related illness | 28 days
  Participant self-report, review of hospital records and discharge summaries within 28 days of randomisation
Pharmacokinetics of favipiravir as measured by Clearance (CL) | Day 7 from randomisation
  Assess pharmacokinetics of favipiravir as measured by Clearance (CL)
Pharmacokinetics of favipiravir as measured by Volume of distribution (V) | Day 7 from randomisation
  Assess pharmacokinetics of favipiravir as measured by Volume of distribution (V)
Pharmacokinetics of favipiravir as measured by Absorption rate constant (Ka) | Day 7 from randomisation
  Assess pharmacokinetics of favipiravir as measured by Absorption rate constant (Ka)
Pharmacokinetics of favipiravir as measured by Maximum concentration (Cmax) | Day 7 from randomisation
  Assess pharmacokinetics of favipiravir as measured by Maximum concentration (Cmax)
Pharmacokinetics of favipiravir as measured by Time to maximum concentration (Tmax) | Day 7 from randomisation
  Assess pharmacokinetics of favipiravir as measured by Time to maximum concentration (Tmax)
Pharmacokinetics of favipiravir as measured by Elimination rate constant (Ke) | Day 7 from randomisation
  Assess pharmacokinetics of favipiravir as measured by Elimination rate constant (Ke)
Pharmacokinetics of favipiravir as measured by Area Under the Curve extrapolated to infinity (AUC (0-inf) | Day 7 from randomisation
  Assess pharmacokinetics of favipiravir as measured by Area Under the Curve extrapolated to infinity (AUC (0-inf)
Pharmacodynamics of favipiravir as measured by Rate of viral load decline (delta) | Day 7 from randomisation
  Assess pharmacodynamics of favipiravir as measured by Rate of viral load decline (delta)
Pharmacodynamics of favipiravir as measured by Maximum increase in viral load under drug treatment (Emax) | Day 7 from randomisation
  Assess pharmacodynamics of favipiravir as measured by Maximum increase in viral load under drug treatment (Emax)
Pharmacodynamics of favipiravir as measured by Concentration to achieve half the maximum possible effect (EC50) | Day 7 from randomisation
  Assess pharmacodynamics of favipiravir as measured by Concentration to achieve half the maximum possible effect (EC50)
Proportion of participants with deleterious or resistance-conferring mutations in SARS-CoV-2 by Day 7 of treatment | Day 7 from randomisation
  Deep sequencing of virus and bioinformatic analysis

CONTACTS AND LOCATIONS:
Overall Officials: David Lowe, Principal Investigator — Institute of Immunity and Transplantation, University College London
Locations (2):
- United Kingdom (2):
  - Royal Free Hospital, London
  - University College London Hospital (UCLH), London

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD has been made at this time.

REFERENCES:
- [Derived] Lowe DM, Brown LK, Chowdhury K, Davey S, Yee P, Ikeji F, Ndoutoumou A, Shah D, Lennon A, Rai A, Agyeman AA, Checkley A, Longley N, Dehbi HM, Freemantle N, Breuer J, Standing JF; FLARE Investigators. Favipiravir, lopinavir-ritonavir, or combination therapy (FLARE): A randomised, double-blind, 2 x 2 factorial placebo-controlled trial of early antiviral therapy in COVID-19. PLoS Med. 2022 Oct 19;19(10):e1004120. doi: 10.1371/journal.pmed.1004120. eCollection 2022 Oct. PMID 36260627
- [Derived] Brown LK, Freemantle N, Breuer J, Dehbi HM, Chowdhury K, Jones G, Ikeji F, Ndoutoumou A, Santhirakumar K, Longley N, Checkley AM, Standing JF, Lowe DM. Early antiviral treatment in outpatients with COVID-19 (FLARE): a structured summary of a study protocol for a randomised controlled trial. Trials. 2021 Mar 8;22(1):193. doi: 10.1186/s13063-021-05139-2. PMID 33685502
- See also: trial results — https://journals.plos.org/plosmedicine/article?id=10.1371/journal.pmed.1004120
- See also: Initial trial Protocol — https://trialsjournal.biomedcentral.com/articles/10.1186/s13063-021-05139-2